CLINICAL TRIAL: NCT02930902
Title: A Preoperative Phase 1B Study to Assess the Safety and the Immunological Effect of Pembrolizumab (Keytruda®) in Combination With Paricalcitol With or Without Chemotherapy in Patients With Resectable Pancreatic Cancer
Brief Title: Pembrolizumab and Paricalcitol With or Without Chemotherapy in Patients With Pancreatic Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0378; NCI-2016-01937 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0378 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Resectable Pancreatic Carcinoma; Stage I Pancreatic Cancer AJCC v6 and v7; Stage IA Pancreatic Cancer AJCC v6 and v7; Stage IB Pancreatic Cancer AJCC v6 and v7; Stage II Pancreatic Cancer AJCC v6 and v7; Stage IIA Pancreatic Cancer AJCC v6 and v7; Stage IIB Pancreatic Cancer AJCC v6 and v7
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; paricalcitol; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (pembrolizumab, paricalcitol) (Active Comparator): Patients receive pembrolizumab IV over 30 minutes on day 1 of each course and paricalcitol IV over 15 minutes on days 1, 8, and 15. Treatment repeats every 21 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Surgical resection is performed within 1 week and up to 4 weeks from last dose of paricalcitol.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paricalcitol; Biological: Pembrolizumab; Procedure: Therapeutic Conventional Surgery
- Arm B (pembrolizumab, paricalcitol, chemotherapy) (Experimental): Patients receive pembrolizumab and paricalcitol as in Arm A. Patients also receive gemcitabine hydrochloride IV over 30 minutes and nab-paclitaxel IV over 30-40 minutes on days 1, 8, and 15 of course 1 in the absence of disease progression or unacceptable toxicity. Surgical resection is performed within 1 week and up to 4 weeks from last dose of paricalcitol.
  Interventions: Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Nab-paclitaxel; Drug: Paricalcitol; Biological: Pembrolizumab; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
  Arms: Arm B (pembrolizumab, paricalcitol, chemotherapy)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
  Arms: Arm B (pembrolizumab, paricalcitol, chemotherapy)
Drug: Paricalcitol — Given IV
  Other Names: Compound 49510; Zemplar
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection of tumor

SUMMARY:
This phase Ib trial studies the side effects and best way to give pembrolizumab and paricalcitol with or without chemotherapy in patients with pancreatic cancer that can be removed by surgery. Monoclonal antibodies, such as pembrolizumab, may find tumor cells and help carry tumor-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab and paricalcitol with or without chemotherapy before surgery may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of neoadjuvant pembrolizumab in combination with paricalcitol with or without gemcitabine and nab-paclitaxel for the treatment of resectable pancreatic cancer.

II. To estimate the number of tumor infiltrating lymphocytes (TILs) in resected pancreatic cancer subjects receiving neoadjuvant pembrolizumab in combination with paricalcitol with or without gemcitabine and nab-paclitaxel.

SECONDARY OBJECTIVES:

I. To estimate the resection rate and pathological response of resectable pancreatic cancer treated with neoadjuvant pembrolizumab in combination with paricalcitol with or without gemcitabine and nab-paclitaxel.

EXPLORATORY CORRELATIVE OBJECTIVES:

I. To estimate the disease free survival (DFS) of resectable pancreatic cancer subjects treated with neoadjuvant pembrolizumab in combination with paricalcitol with or without gemcitabine and nab-paclitaxel.

II. To estimate the overall survival (OS) of subjects with resectable pancreatic cancer who received neoadjuvant pembrolizumab in combination with paricalcitol with or without gemcitabine and nab-paclitaxel.

III. To enumerate CD8+ and CD8+ CD45RO+ cells within and around tumor cell nests, and characterize immunotypes based on distribution of T cells relative to intratumoral vasculature post-neoadjuvant treatment.

IV. To evaluate PD-L1 expression on tumor samples pre- and post-neoadjuvant treatment.

V. To estimate changes in different subsets of T- cells in the peripheral blood pre, during and post-neoadjuvant treatment.

VI. To identify immune signature based on gene expression profiling in tumor samples that may correlate with clinical response in pancreatic cancer patients.

VII. Compare TILs in resected specimen to historical controls of untreated and treated samples.

VIII. To explore the relationship between genomic alterations and treatment administered.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM A: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of each course and paricalcitol IV over 15 minutes on days 1, 8, and 15. Treatment repeats every 21 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Surgical resection is performed within 1 week and up to 4 weeks from last dose of paricalcitol.

ARM B: Patients receive pembrolizumab and paricalcitol as in Arm A. Patients also receive gemcitabine hydrochloride IV over 30 minutes and nab-paclitaxel IV over 30-40 minutes on days 1, 8, and 15 of course 1 in the absence of disease progression or unacceptable toxicity. Surgical resection is performed within 1 week and up to 4 weeks from last dose of paricalcitol.

After completion of study treatment, patients are followed up at 30 days, every 4 months for 1 year, then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial
* Patients must have potentially resectable pancreatic carcinoma and have agreed to undergo surgical resection at Monroe Dunaway (MD) Anderson Cancer Center if operable; they will have undergone staging (physical examination, contrast enhanced computed tomography [CT] or magnetic resonance imaging [MRI] [if CT contraindicated] to determine resectability)
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status 0-1 are eligible
* Have histologically or cytologically confirmed diagnosis of pancreatic carcinoma
* Have no known metastases
* Previous systemic chemotherapy or radiation for pancreatic cancer is not allowed
* In subjects requiring biliary decompression, biliary stent or drainage using percutaneous transhepatic cholangiogram (PTC) are allowed
* Patients must have no fever or evidence of infection or other coexisting medical condition that would preclude administration of study drugs; patients with uncontrolled congestive heart failure, unstable angina and myocardial infarction within 3 months will be excluded
* Have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication, pembrolizumab (cycle 1, day 1) (female subjects of childbearing potential); if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication (male and female subjects of childbearing potential; Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject; acceptable methods of contraception are as follows: single method (one of the following is acceptable): intrauterine device (IUD), vasectomy of a female subject's male partner, contraceptive rod implanted into the skin; combination method (requires use of two of the following): diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide), cervical cap with spermicide (nulliparous women only), contraceptive sponge (nulliparous women only), male condom or female condom (cannot be used together), hormonal contraceptive: oral contraceptive pill (estrogen/progestin pill or progestin-only pill), contraceptive skin patch, vaginal contraceptive ring, or subcutaneous contraceptive injection; abstinence is acceptable if this is the usual lifestyle and preferred contraception method for the subject
* Demonstrate adequate organ function; all screening laboratory tests should be performed within 7 days of treatment initiation
* Patients must have tumor tissue available from a diagnostic or other pre-treatment biopsy of the tumor that is sufficient for tissue analysis as follows:

  * Hematoxylin and eosin (H&E) analysis shows sufficient malignant cell staining of the tissue
  * Formalin-fixed paraffin-embedded (FFPE) cell block that provides a minimum of 10 unstained slides
  * Cell block may be created from multiple-pass fine needle aspiration (FNA) if core needle biopsy (CNB) is not feasible

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy, herbal/complementary oral or IV medicine, or used an investigation device within 4 weeks of the first dose of treatment
* Major cardiovascular or pulmonary comorbidity that precludes use of general anesthesia (NYHA [New York Heart Association] class III and IV)
* Had prior systemic therapy for pancreatic cancer
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment; the use of physiologic doses of corticosteroids may be approved after consultation with the principal investigator (PI) and Merck
* Has a diagnosed additional malignancy within 5 years prior to first dose of study treatment with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected in situ cervical and/or breast cancers
* Has radiographically detectable (even if asymptomatic and/or previously treated) central nervous system (CNS) metastases and/or carcinomatous meningitis as assessed by local site investigator and radiology review
* Has a known history of, or any evidence of, interstitial lung disease or (non-infectious) pneumonitis that required steroids or there is current pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator, including dialysis
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment
* Has received prior immunotherapy including anti-PD-1, anti-PD-L1, or anti-PD-L2 agents, or if the subject has previously participated in Merck pembrolizumab clinical trials
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has documented active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected); in patients without a known history of hepatitis B or C, serologies should be obtained at screening
* Has received a live vaccine within 30 days of planned start of study therapy (cycle 1, day 1); Note: the killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* Has laboratory evidence of hypercalcemia (>= 11 mg/dl [in presence of normal albumin]) and/or hyperphosphatemia (>= 5.5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicities as defined by Common Terminology Criteria for Adverse Events version 4.0 | Up to 11 weeks
  Incidence will be descriptive.

SECONDARY OUTCOMES:
Resection rate | Up to 7 weeks (within 1 week of end of neoadjuvant treatment)
  Summary statistics will be used.

OTHER OUTCOMES:
Disease free survival (DFS) | Up to 3 years
  The analysis will be descriptive only. Summary statistics estimated using the Kaplan-Meier method.
Overall survival (OS) | Up to 3 years
  The analysis will be descriptive only. Summary statistics estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon G Smaglo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org